CLINICAL TRIAL: NCT07380984
Title: A Prospective Study to Evaluate the Efficacy and Safety of PD-1 Monoclonal Antibody-based Stratified Targeted Therapy Combined With Concurrent Radiotherapy for Patients With Treatment-naive Early-stage Nasal-type NK/T-cell Lymphoma
Brief Title: PD-1 Antibody-based Therapy With Concurrent RT for Early-stage NKTCL
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Zhao Weili, Professor and Director，Shanghai Institute of Hematology, Ruijin Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NOVEL-01
Record Dates: First submitted 2026-01-24; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Natural Killer/T-cell Lymphoma
MeSH Terms: interventions — spartalizumab; Radiotherapy; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PD-1 antibody monotherapy group (Experimental): Patients will receive concurrent standard involved-site radiotherapy (ISRT) and PD-1 monoclonal antibody therapy. Administration of PD-1 mAb will start on Day 1 of radiotherapy (C1D1) at a dose of 200 mg via intravenous infusion over 30 minutes or longer, once every 3 weeks. After the 3rd cycle, patients will undergo re-evaluation (PET scan and plasma EBV DNA detection). Patients with an interim Deauville score of 1-3 and negative EBV DNA will continue to receive 3 cycles of PD-1 monoclonal antibody therapy.
  Interventions: Drug: PD-1 antibody; Radiation: radiotherapy
- The multi-drug combination group (Experimental): Patients will receive concurrent standard involved-site radiotherapy (ISRT) and PD-1 monoclonal antibody therapy. Administration of PD-1 mAb will start on Day 1 of radiotherapy (C1D1) at a dose of 200 mg via intravenous infusion over 30 minutes or longer, once every 3 weeks. After the 3rd cycle, patients will undergo re-evaluation (PET scan and plasma EBV DNA detection). Patients with an interim Deauville score of 4-5 or positive EBV DNA will subsequently receive 3 cycles of a combination regimen of PD-1 antibody, chidamide and golidocitinib.
  Interventions: Drug: PD-1 antibody; Radiation: radiotherapy; Drug: Chidamide; Drug: golidocitinib

INTERVENTIONS:
Drug: PD-1 antibody — Administration of PD-1 mAb will start on Day 1 of radiotherapy (C1D1) at a dose of 200 mg via intravenous infusion over 30 minutes or longer, once every 3 weeks, cycle 1 - cycle 6
Radiation: radiotherapy — Concurrent standard involved-site radiotherapy (ISRT)
Drug: Chidamide — The dosage of chidamide will follow a dose-escalation design: 20 mg twice weekly (biw) in the first stage, then escalated to 30 mg biw, using the Bayesian Optimal Interval (BOIN) design to determine the recommended dose, followed by dose expansion in the second stage, every 3 weeks, cycle 4 - cycle 6.
  Arms: The multi-drug combination group
Drug: golidocitinib — Golidocitinib will be administered at a dose of 150 mg once daily (qd), every 3 weeks, cycle 4 - cycle 6.
  Arms: The multi-drug combination group

SUMMARY:
Natural killer/T-cell lymphoma (nasal type) is a mature T/NK-cell lymphoma closely associated with Epstein-Barr virus (EBV), with a high prevalence among populations in Asia and South America. It primarily occurs at extranodal sites, including the nasal/paranasal regions, skin, gastrointestinal tract, and other organs. This study focuses on previously untreated patients with early-stage NKTCL (nasal type), exploring a response-adapted comprehensive therapeutic strategy that combines PD-1 monoclonal antibody-based stratified targeted therapy with concurrent radiotherapy. The aim is to provide integrated management for early-stage extranodal NK/T-cell lymphoma (nasal type), and reduce toxicity while improving overall treatment outcomes for patients.

ELIGIBILITY:
Inclusion Criteria:

* The subject has histopathologically confirmed extranodal NK/T-cell lymphoma, nasal type (according to the 2022 WHO classification).
* No prior history of anti-lymphoma therapy.
* Age ≥ 18 years.
* Life expectancy > 3 months.
* Ann Arbor stage I-II.
* At least one measurable/evaluable disease site confirmed by diagnostic biopsy prior to the initiation of treatment.
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2.
* Signed informed consent form (ICF).
* Willingness and ability to comply with the study protocol.
* Sufficient bone marrow, hepatic, and renal function, defined as:

  1. Absolute neutrophil count (ANC) > 1,000/μL
  2. Platelet count > 50,000/μL
  3. Hemoglobin > 9 g/dL
  4. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 3× upper limit of normal (ULN)
  5. Serum total bilirubin < 1.5 × ULN (patients with Gilbert's syndrome are eligible)
  6. Serum creatinine < 2 × ULN or creatinine clearance > 50 mL/min
* Availability of tumor tissue samples (preferably fresh tissue; archived tissue samples are acceptable).
* For women of childbearing potential, agreement to use adequate contraception to avoid pregnancy during the study treatment period.
* For male, agreement to remain abstinent or use a barrier method of contraception.

Exclusion Criteria:

* Advanced-stage disease (Ann Arbor Stage III-IV).
* Nonnasal-type NKTCL.
* A history of autoimmune disease requiring systemic treatment (i.e., with disease-modifying antirheumatic drugs, corticosteroids, or immunosuppressants) within the past 2 years, including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody-associated vasculopathy, granulomatosis with polyangiitis (Wegener's), Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.

The following conditions are permissible for enrollment: patients with autoimmune hypothyroidism or type 1 diabetes receiving stable treatment; hormone replacement therapy (e.g., levothyroxine, insulin, or supplementation with physiological hormones for adrenal or pituitary insufficiency) is not considered systemic therapy and is allowed.

* A history of other invasive malignancies within the past 3 years that has not been treated with curative intent or is currently receiving anticancer therapy (including hormonal therapy for breast or prostate cancer).
* A history of (non-infectious) pneumonia requiring corticosteroid therapy; or clinical evidence of interstitial lung disease or active, non-infectious pneumonia.
* Active infections requiring systemic treatment, including:

  1. A known history of active tuberculosis;
  2. Positive results for HBsAg, HCV, or HIV; HBV seropositivity is permitted only if HBV DNA < 1000 IU/mL;
  3. Active viral infections other than hepatitis B and C (e.g., herpes zoster).
* Severe cardiovascular disease, including myocardial infarction, unstable arrhythmia, or unstable angina occurring within the past 3 months.
* Prior treatment with anti-PD-1, anti-PD-L1, or anti-PD-L2 agents.
* Administration of live-attenuated vaccines within 4 weeks prior to the initiation of study treatment; patients are prohibited from receiving live-attenuated vaccines during the study period, including influenza vaccines.
* Use of systemic immunosuppressive agents within 2 weeks prior to the initiation of study treatment, or planned use of such agents during the study period, including cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor (anti-TNF) drugs.
* Evidence of central nervous system involvement.
* A history of allogeneic tissue/solid organ transplantation.
* A history of severe hypersensitivity reactions (Grade ≥ 3) to PD-1 monoclonal antibodies and/or their excipients, or to gorlitinib and/or its excipients.
* Any other factors judged by the investigator to potentially affect compliance with the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-02-01 (Estimated); Study Completion 2029-02-01 (Estimated)

PRIMARY OUTCOMES:
2-year progression-free survival rate | Baseline up to data cut-off (up to 24 months).
  Progression-free survival is defined as the time from registration to the first occurrence of disease progression or relapse, using 2014 Lugano criteria, or death from any cause. For patients who received subsequent treatment after the interim assessment, the endpoint shall be defined by the event first occurring after the initiation of subsequent treatment.

SECONDARY OUTCOMES:
Complete Response Rate | At the end of cycle 3, cycle 6 after treatment start.
  The proportion of patients with complete response after 3 cycles, 6 cycles from treatment start, according to the 2014 Lugano Response Criteria.
Overall Response Rate | At the end of cycle 3, cycle 6 after treatment start.
  The proportion of patients with complete and partial response after 3 cycles, 6 cycles from treatment start, according to the 2014 Lugano Response Criteria.
2-year overall survival rate | Baseline up to data cut-off (up to 24 months).
  Overall survival is defined as the time from registration to death from any cause.
2-year event-free survival rate | Baseline up to data cut-off (up to 24 months).
  Event-free survival is defined as the time from registration to event occurrence. An event is defined as one of the following: disease progression, death from any cause, discontinuation of the protocol-specified treatment due to adverse events, or initiation of a new anti-lymphoma therapy.
Duration of Response | From enrollment to study completion (up to approximately 24 months).
  Duration of response is defined as the period from the first response to first evidence of disease progression, relapse or death of any cause.
Treatment-Related Adverse Events rate | From enrollment to study completion (up to approximately 24 months).
  Adverse events will be graded by the investigator according to the NCI-CTCAE Version 5.0.
The change of plasma EB virus DNA load | Baseline up to data cut-off (up to 24 months).
  The change of plasma EB virus DNA load during the treatment